CLINICAL TRIAL: NCT06917209
Title: Evaluation of the Efficacy of Dissociation-Focused Cognitive Behavior Therapy: a Multicenter Randomized Controlled Trial
Brief Title: Evaluation of the Efficacy of Dissociation-Focused Cognitive Behavior Therapy
Acronym: TCC-DISSO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR240330
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Dissociative Disorder
MeSH Terms: conditions — Dissociative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group will receive 9 weekly sessions of DF-CBT psychotherapy. (Experimental)
  Interventions: Other: CBT-CD psychotherapy
- The control group will receive 9 weekly relaxation sessions. (No Intervention)

INTERVENTIONS:
Other: CBT-CD psychotherapy — 9 weekly sessions of CBT-CD psychotherapy
  Arms: The experimental group will receive 9 weekly sessions of DF-CBT psychotherapy.

SUMMARY:
Dissociative symptoms and disorders are particularly prevalent in the general population and among people suffering from psychiatric disorders. To date, no treatment has proven effective for this type of problem. Exploratory studies (without control group) have been carried out. Among these studies, dissociation-focused cognitive behavioral therapy (DF-CBT) seems promising. DF-CBT is based on a solid empirical model that has received numerous scientific evidence.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Membership of a social security scheme
* Participant's express consent
* Have at least one diagnosis of dissociative disorder among the following:

depersonalization/derealization disorder, dissociative identity disorder, unspecified dissociative disorder.

* Be able to carry out psychotherapy sessions.
* If taking psychiatric medication, treatment must have been stable for at least 30 days.

Exclusion Criteria:

* Present one of the following current diagnoses: substance use disorder (excluding tobacco), neurodevelopmental disorder, anorexia nervosa, severe depressive disorder, schizophrenia spectrum disorder, bipolar disorder, personality disorder other than borderline personality disorder.
* Present cognitive deficits.
* Be engaged in psychotherapeutic work.
* Be undergoing benzodiazepine treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2027-05-22 (Estimated)

PRIMARY OUTCOMES:
Difference in Dissociative Experience Scale (DES) | Between randomization and 3 months after
  Difference in Dissociative Experience Scale (DES) between randomization and 3 months after.
  The DES assesses dissociation through 28 items. The total score ranges between 0 and 100, where high scores indicate high levels of dissociation.

SECONDARY OUTCOMES:
Hetero-administered visual analogue scale | At randomization, 3 months and 6 months after
  Visual analogue scales in which the practitioner rates the intensity of the patient's dissociative symptoms on the basis of his/her clinical assessment.
Dissociation Questionnaire (DIS-Q) | At randomisation, 3 months and 6 months after
  The Dissociation Questionnaire is a 63-item questionnaire measuring dissociative-trait manifestations. Participants respond to each item using a 5-point Likert scale. Four sub-scores (loss of control, absorption, amnesia and identity confusion) are calculated.
Hospital Anxiety Depression Scale (HADS) | Randomization, 3 months and 6 months after
  Hospital Anxiety Depression Scale (HADS) is a 14-item self-report questionnaire. Two sub-scores (anxiety and depression) are calculating.
  Both scores range between 0 and 21 with 0 corresponding to the ideal score (no anxiety or depression symptoms).
Post traumatic stress disorder checklist scale (PCL-5) | Randomization, 3 months and 6 months after
  The post traumatic stress disorder checklist scale (PLC-5) is 20-item scale to assess post-traumatic stress symptoms. Participants respond to each item using a 5-point Likert scale. The score ranges between 0 and 80, with 0 reflecting no post traumatic stress disorder.
Satisfaction With Life Scale (SWLS) | Randomization, 3 months and 6 months after
  The Satisfaction With Life Scale (SWLS) is a 5-item questionnaire assessing quality of life. Participants respond to each item using a 7-point Likert scale. The score range bewteen 0 and 35 with 35 reflects an extreme satisfaction with life.
Dissociative Experiences Scale (DES) | At 6 months after randomization
  The DES assesses dissociation through 28 items. The total score ranges between 0 and 100, where high scores indicate high levels of dissociation.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis VANCAPPEL, PhD, Study Chair — Clinique Psychiatrique Universitaire / CHRU de Tours; Wissam EL HAGE, MD-PhD, Principal Investigator — Clinique Psychiatrique Universitaire CPU / CHRU de Tours
Locations (8):
- France (8):
  - Psychiatrie / CHU ANGERS, Angers
  - Centre régional du Psychotraumatisme des Hauts de France / CHU LILLE, Lille
  - Urgences psychiatrique / CHU MONTPELLIER, Montpellier
  - Unité de neuromodulation en psychiatrie / CHU NANTES, Nantes
  - Centre départemental de Psychotraumatologie (unité TCC) / ORLEANS, Orléans
  - Centre Régional du Psychotraumatisme du Grand Est / CHU STRASBOURG, Strasbourg
  - Centre Régional du Psychotraumatisme CRP / CHRU TOURS, Tours
  - Clinique Psychiatrique Universitaire / CHRU de Tours, Tours